CLINICAL TRIAL: NCT05771298
Title: Potassium Titanyl Phosphate Laser Versus Pulsed Dye Laser for Rosacea - a Prospective Case-Control Study
Brief Title: Potassium Titanyl Phosphate Laser Versus Pulsed Dye Laser for Rosacea - a Prospective Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-22
Record Dates: First submitted 2023-03-05; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potassium Titanyle Phosphate (KTP) Laser (Other): Subjects will be treated with a KTP laser in 1 - 3 sessions at intervals of 4 - 6 weeks.
  Interventions: Device: 532nm KTP
- Pulsed Dye Laser (Other): Subjects will be treated with a PDL in 1 - 3 sessions at intervals of 4 - 6 weeks.
  Interventions: Device: 585nm PDL

INTERVENTIONS:
Device: 532nm KTP — one to three treatment sessions
  Arms: Potassium Titanyle Phosphate (KTP) Laser
Device: 585nm PDL — one to three treatment sessions
  Arms: Pulsed Dye Laser

SUMMARY:
To compare the efficacy and safety of 532 nm KTP and 585 nm PDL for treating rosacea.

DETAILED DESCRIPTION:
Rosacea is a common, chronic inflammatory skin disease that usually affects the cheeks, nose, forehead, and chin [1]. Clinically, it presents initially with transient erythema (flushing) and telangiectasia. As it progresses, persistent erythema and papules and pustules appear. Phymatous changes result from hypertrophy of the sebaceous glands, and usually manifest as rhinophyma, gnatophyma, and metophyma [2]. Depending on the literature, rosacea has a prevalence of 1% to 22% [3]. Time of manifestation of the disease is usually between 30 and 50 years [4]. Women are more frequently affected [4].

For laser treatment of rosacea, the pulsed dye laser (PDL) with a wavelength of 595nm is frequently used. The treatment includes at least three sessions at intervals of about 4 weeks and leads to lightening and reduction of the lesions as well as reduction of papules and pustules. Various clinical studies have already demonstrated the high efficacy of PDL [5-7]. The treatment is painless, and local or general anesthesia is not necessary.

The KTP laser is also an option in the treatment of rosacea. Due to the more stable technology of the frequency-doubled Nd:YAG (KTP) and associated lower maintenance problems, this laser system appears to be a safer and more reliable treatment option for rosacea patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years and older
* Good general health, no relevant previous diseases
* Presence of rosacea
* Cognitive ability and willingness to give consent (Informed Consent)

Exclusion Criteria:

* Age < 18 years
* Pregnant and breastfeeding women
* Significant open wounds or lesions of the region to be treated
* Metallic implants in the region to be treated
* Missing consent and/or data protection declarations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
reduction of erythema | at follow-up visit 4 weeks after last treatment session
  assessment scale 0 - 4 (normal skin - severe erythema) evaluated by physician and blinded investigator
pain intensity | at follow-up visit 4 weeks after last treatment session
  using numeric rating scale 0 - 10 (none - unbearable pain) evaluated by subjects
swelling | at follow-up visit 4 weeks after last treatment session
  assessment scale 1 - 6 (very - none) evaluated by subjects
purpura | at follow-up visit 4 weeks after last treatment session
  assessment scale 1 - 6 (very - none) evaluated by subjects

SECONDARY OUTCOMES:
patient satisfaction | at follow-up visit 4 weeks after last treatment session
  assessment scale 1 - 6 (very - not at all) evaluated by subjects

CONTACTS AND LOCATIONS:
Overall Officials: L Nguyen, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Laser Department, University Medical-Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Zuuren EJ, Fedorowicz Z, Carter B, van der Linden MM, Charland L. Interventions for rosacea. Cochrane Database Syst Rev. 2015 Apr 28;2015(4):CD003262. doi: 10.1002/14651858.CD003262.pub5. PMID 25919144
- [Background] van Zuuren EJ. Rosacea. N Engl J Med. 2017 Nov 2;377(18):1754-1764. doi: 10.1056/NEJMcp1506630. No abstract available. PMID 29091565
- [Background] Tan J, Berg M. Rosacea: current state of epidemiology. J Am Acad Dermatol. 2013 Dec;69(6 Suppl 1):S27-35. doi: 10.1016/j.jaad.2013.04.043. PMID 24229634
- [Background] Elewski BE, Draelos Z, Dreno B, Jansen T, Layton A, Picardo M. Rosacea - global diversity and optimized outcome: proposed international consensus from the Rosacea International Expert Group. J Eur Acad Dermatol Venereol. 2011 Feb;25(2):188-200. doi: 10.1111/j.1468-3083.2010.03751.x. Epub 2010 Jun 25. PMID 20586834
- [Background] Kim BY, Moon HR, Ryu HJ. Comparative efficacy of short-pulsed intense pulsed light and pulsed dye laser to treat rosacea. J Cosmet Laser Ther. 2019 Aug;21(5):291-296. doi: 10.1080/14764172.2018.1528371. Epub 2018 Oct 4. PMID 30285506
- [Background] Osman M, Shokeir HA, Hassan AM, Atef Khalifa M. Pulsed dye laser alone versus its combination with topical ivermectin 1% in treatment of Rosacea: a randomized comparative study. J Dermatolog Treat. 2022 Feb;33(1):184-190. doi: 10.1080/09546634.2020.1737636. Epub 2020 Mar 12. PMID 32141785
- [Background] Bernstein EF, Schomacker K, Paranjape A, Jones CJ. Pulsed dye laser treatment of rosacea using a novel 15 mm diameter treatment beam. Lasers Surg Med. 2018 Oct;50(8):808-812. doi: 10.1002/lsm.22819. Epub 2018 Apr 10. PMID 29635699
- [Derived] Nguyen L, Seeber N, Kautz G, Hartjen A, Schneider SW, Herberger K. 532-nm potassium titanyl-phosphate laser versus 595-nm pulsed dye laser for port-wine birthmarks: A prospective, randomized, split-side study. J Eur Acad Dermatol Venereol. 2024 Jun;38(6):1140-1146. doi: 10.1111/jdv.19750. Epub 2023 Dec 21. PMID 38794945